CLINICAL TRIAL: NCT05750771
Title: Comparison of Drug-coated Balloon and Drug-eluting Stent for Severe Calcification of de Novo Lesion in Elderly Coronary Heart Disease
Brief Title: Comparison of DCB and DES for Severe Calcification of de Novo Lesion in Elderly CHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE202303
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB Group (Experimental): Implantation of drug-coated balloons in patients with satisfactory pretreatment
  Interventions: Device: DCB
- DES Group (Experimental): Implantation of drug-eluting stents in patients with satisfactory pretreatment
  Interventions: Device: DES

INTERVENTIONS:
Device: DES — Second-generation drug-eluting stents
  Arms: DES Group
Device: DCB — Drug-coated balloon with paclitaxel as drug coating
  Arms: DCB Group

SUMMARY:
The goal of this clinical trial was to compare the effectiveness of drug balloons versus drug-coated stents in calcified lesions in elderly coronary artery disease. The main question it aims to answer is whether the application of DCB is non-inferior to DES for in situ large vessel calcified lesions in the elderly coronary arteries.

And to develop a method to precisely identify the nature and extent of calcified lesions and to rationalize the choice of pretreatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. older than 60 years of age.
* 2. meeting the indications for coronary intervention.
* 3. IVUS examination suggests severe calcified lesions (calcification angle > 270° at the target lesion) or OCT examination suggests severe calcified lesions (calcification angle > 180° and/or length > 5 mm and/or thickness > 0.5 mm);
* 4. Target lesion vessel diameter > 2.5 mm

Exclusion Criteria:

* 1. inability to provide written informed consent.
* 2. unable to administer antiplatelet agents and anticoagulant therapy; have allergies to heparin, contrast agents, etc.
* 3. the subject is participating in another uncompleted clinical trial
* 4. life expectancy <1 year.
* 5. non-in situ vascular lesions.
* 6. cardiogenic shock.
* 7. Patients with hemodynamic instability

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
LLL | 12 months
  Late lumen loss (LLL) of the target lesion segment

SECONDARY OUTCOMES:
MACE | Perioperative period, 30 days, 3 months, 6 months, 12 months after discharge
  Cardiovascular death, target vessel revascularization, target vessel non-lethal myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — Fuwai central China cardiovascular hospotial
Locations (1):
- Fuwai central China cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No